CLINICAL TRIAL: NCT06111638
Title: A Study to Evaluate the Safety, Tolerability and Efficacy of an Adeno-associated Viral Vector Containing an Expression Cassette of the Human Factor VIII Transgene (BBM-H803) Injection in Participants With Hemophilia A
Brief Title: Evaluation of the Safety and Efficacy of Hemophilia A Gene Therapy Drugs
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Xinzhi BioMed Co., Ltd. (Industry)
Collaborators: Shanghai MYGT Biopharmaceutical LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBM002-CLN1001
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; gene therapy; Adeno-Associated Virus
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm of BBM-H803 (Experimental): The dose of BBM-H803 will be calculated according to participant's weight
  Interventions: Genetic: Single dose intravenous injection of BBM-H803

INTERVENTIONS:
Genetic: Single dose intravenous injection of BBM-H803 — Single dose intravenous infusion of BBM-H803, an adeno-associated viral (AAV) vector derived from recombinant DNA techniques to contain an expression cassette of the human factor VIII transgene in liver. The dose of BBM-H803 will be calculated according to participant's weight.

SUMMARY:
This is a multi-center, single-arm, open-label, single-dose treatment clinical study to evaluate the safety, tolerability and efficacy of BBM-H803 injection in severe Hemophilia A subjects.

BBM-H803 is an adeno-associated viral (AAV) vector derived from recombinant DNA techniques to contain an expression cassette of the human factor VIII transgene and raises circulating levels of endogenous FVIII.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily sign informed consent form;
2. Males ≥ 18 years;
3. Subjects are clinically diagnosed with severe hemophilia A;
4. Have > = 150 documented exposure days to a Factor VIII protein product
5. No prior history of hypersensitivity or anaphylaxis associated with any FVIII immunoglobulin;
6. Use a reliable contraception method during the study;
7. Capsid antibody negative;
8. Subjects have good compliance.

Exclusion Criteria:

1. Being positive for hepatitis B surface antigen (HBsAg) or hepatitis B virus-DNA (HBV-DNA). Being positive for hepatitis C virus antibody (HCV-Ab) or hepatitis C virus RNA (HCV-RNA).

   Subjects with medical history of hepatitis B or C can be regarded as negative only when 2 required samplings are conducted at least 3 months apart and both test results of indicators aforementioned are negative, HIV positive patients or Syphilis seropositive patients;
2. Currently on antiviral therapy for hepatitis B or C;
3. Suffer from coagulation disorders other than hemophilia A;
4. In addition to glucocorticoids, any other immunosuppressants are being used before selection;
5. Have vaccination history within 2 months before administration, or vaccination schedule during immunomodulatory therapy;
6. Have potential liver diseases, such as previous diagnosis of portal hypertension, splenomegaly, hepatic encephalopathy or liver fibrosis (fibrosis stage ≥ 3); nodules or cysts were found by B ultrasound, or elevated alpha-fetoprotein was detected by laboratory tests. Subjects who are not eligible for the study if the abnormalities are clinically significant regarding to the medical judgement of the investigator;
7. Scheduling of elective major surgery known or planned during the insertion period or the 52-week study period following BBM-H803 infusion;
8. Have participated in a previous gene therapy research trial before screening or have used other test drugs within 4 weeks before screening, or within 5 half-life of the test drug, whichever is longer; Have received emesezumab within 6 months before screening; Or drugs evaluated by the researcher to affect the study;
9. Any herbal preparations (herbal supplements or traditional Chinese medicines of plant, mineral or animal origin) used during the 4 weeks prior to or during the study that may affect liver function, except topical use; Or any Chinese herbal medicine that the researcher evaluates to affect the study;
10. Have alcohol or drug addiction, or cannot stop drinking as advised by the researcher throughout the study;
11. Have acute/chronic infections or other chronic diseases that may pose a risk for the study, or have a major illness, who have a current or previous history of malignant tumors, or who have other unstable medical conditions, including poor mental state and risk of suicide, that the investigator deems unsuitable for participation in the study;
12. Any other conditions that the investigator deems unsuitable for participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) events | 6 weeks
  To access the numbers of DLT events determined by the Safety Data Review Committee (SRC) in DLT observation period after BBM-H803 injection infusion
The incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | 6 weeks
  To assess the safety of BBM-H803 Injection by TEAEs and SAEs.
Number of participants with Changes in liver function | 6 weeks
  To assess changes in liver function before and after treatment, including alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), alkaline phosphatase (ALP), and gamma-glutamyl transpeptidase (GGT)

SECONDARY OUTCOMES:
Plasma FVIII activity level | 52 weeks
  All samples collected from participants for plasma FVIII activity levels were analyzed and used to determine peak and steady-state vector-derived circulating FVIII activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Study Chair — Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (8):
- China (8):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Southern Hospital, Southern Medical University, Guangzhou, Guangdong
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Wuhan Union Hospital Affiliated to Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No